CLINICAL TRIAL: NCT04494022
Title: Role of Sonazoid-enhanced Ultrasound as a Secondary Diagnostic Modality in Non-invasive Diagnostic Algorithms for Hepatocellular Carcinoma
Brief Title: Role of CEUS as a Secondary Diagnostic Modality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Pf., Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2004-035-1116
Record Dates: First submitted 2020-06-05; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: All participants underwent CEUS. The image reviews based on cross-section images will be performed with or without CEUS results. Two image sets (cross-sectional image with CEUS and without CEUS) will be compared.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cross-sectional image only (No Intervention): Image set which consists of a Cross-sectional image only.
- Cross-sectional image with CEUS (Active Comparator): The same participants with Arm1. But image set will consist of a Cross-sectional image and CEUS.
  Interventions: Diagnostic Test: contrast enhanced ultrasound

INTERVENTIONS:
Diagnostic Test: contrast enhanced ultrasound — Perflubutane enhanced ultrasound for evaluating hepatic tumor
  Arms: Cross-sectional image with CEUS

SUMMARY:
To determine the role of contrast-enhanced ultrasound (CEUS) as a second-line imaging modality after gadoxetate-enhanced MRI (Gd-EOB-MRI) for identifying hepatocellular carcinoma (HCC) among at-risks observations.

DETAILED DESCRIPTION:
The purpose of our study was to evaluate the diagnostic ability of CEUS with perflubutane to identify HCC on the indeterminate observation in Gd-EOB-MRI and to establish the role of CEUS as a second-line (post-Gd-EOB-MRI) modality for HCC diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* at risk of HCC by Liver Imaging Reporting and Data System (LI-RADS)
* at least one treatment-naïve solid hepatic observation (≥1 cm) while surveillance using US, CT or MRI
* signed informed consent

Exclusion Criteria:

* congestive hepatopathies
* severe cardiovascular dysfunction
* no recent cross-sectional images within 4 weeks
* suboptimal cross-sectional images quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Compared the image features of CEUS and Gd-EOB-MRI in at-risk observation | 1. For 3 days after undergoing CEUS to check the complication of CEUS, per each participants. 2. The time interval between CEUS and Gd-EOB-MRI should not be exceed 4 weeks.
  Compared the frequency of arterial phase hyperenhancement (APHE) and washout in at-risk observation, between CEUS and Gd-EOB-MRI.
Compared diagnostic performance of Gd-EOB-MRI alone and Gd-EOB-MRI with CEUS. | 1. For 3 days after undergoing CEUS to check the complication of CEUS, per each participants. 2. The time interval between CEUS and Gd-EOB-MRI should not be exceed 4 weeks.
  Evaluated sensitivity, specificity and accuracy for diagnose HCC by using Gd-EOB-MRI alone, or Gd-EOB-MRI with CEUS.

SECONDARY OUTCOMES:
Comparing image characters between two types of ultrasound contrast media | For 3 days after undergoing CEUS to check the complication of CEUS, per each participants.
  Comparing image characters between two types of ultrasound contrast media

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, M.D., Study Director — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: For two years after publication.
Access Criteria: except you want to use illegal purpose